CLINICAL TRIAL: NCT05767073
Title: LIVES: Development of/a Personalized Lifestyle Intervention for Patients With Depression in Psychiatric Outpatient Care and General Practice in a Pilot Study
Brief Title: LIVES: Personalized Lifestyle Intervention for Patients With Depression
Acronym: LIVES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: GGZ Drenthe Mental Health Institution (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11178
Record Dates: First submitted 2022-12-16; First posted 2023-03-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Risk; Depression, Unipolar; Depression, Bipolar
Keywords: depression; lifestyle; mental health care; general practice
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Un controlled cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Lifestyle intervention
  Interventions: Behavioral: Lifestyle InterVEntion (LIVE)

INTERVENTIONS:
Behavioral: Lifestyle InterVEntion (LIVE) — The lifestyle intervention Coaching on Lifestyle (CooL) (van Rinsum 2018)),formed the basis of LIVE and was adapted to specific dysfunctional elements in depressed patients regarding motivation and self-management.
  The focus is on reducing depressive symptoms, enhancing the quality of life and possibly achieving weight loss.
  The lifestyle intervention lasts six months, with 13 weekly 1.5 to 2 hour group sessions and five 45 to 60 -minute individual sessions with at least one person from the patient's support network of friends or family (preferably sharing the same household). All sessions end with individual homework exercises, and each session starts with a 10 to 15-minute positive psychology intervention (PPI) and 5 to 15 minutes of physical activity. These sessions are followed by two booster sessions after about two and six months. Groups consist of 4-8 people.

SUMMARY:
Persons with affective disorder have a considerably increased risk of cardiovascular disease. To a considerable extent, this is due to an unhealthy life style. At present, no adequate lifestyle interventions are available for these patients. In the present pilot intervention study we study the acceptability and feasibility of a newly developed lifestyle intervention that is specifically tailored to the needs of patients with affective disorders treated in mental health care or general practice.

DETAILED DESCRIPTION:
Rationale: Patients with bipolar disorder and severe depressions have a 10-year shorter life expectancy, on average, than the population as a whole. Also patients with less severe depression are still at a substantially increased risk of cardiovascular events. This may be attributed primarily to somatic complications resulting from a largely sedentary existence and an unhealthy lifestyle related to their disorder and/or the side effects of psychopharmacological treatment. Generally speaking, multimodal lifestyle interventions are about as effective as medication in reducing cardiovascular risks. Very little research has been conducted into the effect of lifestyle interventions among outpatients in mental health care or patients with mental health problems in general practice. This study seeks to examine the extent to which a personalised lifestyle approach can promote the physical health and quality of life of outpatients and general practice patients with affective disorders.

Objective: The objective of this study is to develop a personalised state-of-the art lifestyle intervention that is both feasible and acceptable to outpatients with bipolar and severe recurrent depressive disorder and to patients with depression in general practice Study design: An explorative pilot study (n = 38) with baseline measurement and different follow-up measurements during and after the intervention.

Study population: Patients (18-65 years old) with bipolar disorder or severe recurrent depression who are being treated at GGZ Drenthe (N=30) and patients with depression in primary care (N=8).

Intervention (if applicable): A personalised multimodal lifestyle intervention consisting of several modules comprising both individual and group sessions. The support network is involved during the individual sessions.

Main study parameters/endpoints: Feasibility and acceptability of the lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

For patients in mental health care only:

* Outpatients
* Diagnosed during intake, the primary diagnosis being chronic bipolar disorder (type I or 2) or a chronic or recurrent severe depression in the narrower sense of the word
* Receiving psychopharmacological treatment
* Have had a physical and lifestyle Routine Outcome Monitoring measurement showing that three or more metabolic parameters were outside the normal range

For patients in general practice (GP) only:

* Diagnosis of depressive symptoms or depressive disorder in the past year as registered in the general practice electronic health record and coded according to the International Classification of Primary Care (ICPC) as P03 and P76, respectively,
* At least mild depressive symptom level according to the Beck Depression Inventory-II (BDI) (score ≥14)
* Body mass index ≥ 25 kg/m2 or increased waist circumference (>88cm (women) of >102cm (men)).

For both patient groups:

- 18 years or older and capable to participate in the intervention according to the treating physician Availability of one or two people close to the patient (friends or family, preferably sharing the same household), i.e. to act as the buddy of the patient.

Exclusion Criteria:

* For GP patients only: current treatment in mental health care (GGZ in Dutch)
* For GP patients only: severe somatic / neurological disease at the discretion of the GP
* Currently participating in another lifestyle intervention
* Insufficient proficiency in Dutch
* Unability to read and write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Reach of LIVE | 27 months (September 2020 through November 2022)
  Reach of our intervention as defined by the absolute number, proportion, and representativeness of individuals who are willing to participate in LIVE
Adherence to LIVE | 18 weeks
  Adherence to the LIVE lifestyle intervention as defined by the number of sessions attended by the participant out of the total of 18 sessions
Drop out from LIVE | 18 weeks
  Drop-out from the LIVE intervention as defined by the proportion of participants who decide to prematurely stop taking part in the LIVE intervention
Feasibility and acceptability of the LIVE intervention according to the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 3
  Feasibility and acceptability of the LIVE intervention will be assessed using qualitative interviews Participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 6
  Feasibility and acceptability of the LIVE intervention will be assessed using qualitative interviews Participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 9
  Feasibility and acceptability of the LIVE intervention will be assessed using qualitative interviews Participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 12
  Feasibility and acceptability of the LIVE intervention will be assessed using qualitative interviews Participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 15
  Feasibility and acceptability of the LIVE intervention will be assessed using qualitative interviews Participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 18
  Feasibility and acceptability of the LIVE intervention will be assessed using qualitative interviews Participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed

SECONDARY OUTCOMES:
Feasibility and acceptability of the LIVE intervention according to the buddy of the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 3
  Feasibility and acceptability will be assessed using qualitative interviews. Buddies of participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the buddy of the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 6
  Feasibility and acceptability will be assessed using qualitative interviews. Buddies of participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the buddy of the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 9
  Feasibility and acceptability will be assessed using qualitative interviews. Buddies of participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the buddy of the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 12
  Feasibility and acceptability will be assessed using qualitative interviews. Buddies of participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the buddy of the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 15
  Feasibility and acceptability will be assessed using qualitative interviews. Buddies of participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Feasibility and acceptability of the LIVE intervention according to the buddy of the participant as assessed by qualitative interviews and qualitative data analysis | Up to week 18
  Feasibility and acceptability will be assessed using qualitative interviews. Buddies of participants will be interrogated on how they experienced themes during the different modules of the intervention. A topic-list will be used by the interviewer to check whether all relevant themes on feasibility and acceptability have been discussed
Quality of life as assessed by The Manchester Short Assessment of Quality of Life (MANSA). | Baseline, at the end of the intervention 18 weeks after baseline, and at the 6 months follow up (42 weeks after baseline)
  The MANSA measures quality of life focusing on satisfaction with life as a whole and with life domains and consists of a 12-item self-report questionnaire
Depressive symptoms according to the Beck Depression Inventory-II (BDI-II) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The BDI-II is a self-report (21 items) rating inventory which measures depressive symptom level
Recovery of the participant according to the Individual Recovery Outcomes Counter (I.ROC) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The I.ROC is an instrument to quantitatively measure recovery. It uses three indicators on four areas of wellbeing, namely home, opportunity, people, empowerment.
Wellbeing as assessed by the Mental Health Continuum Short Form (MHC-SF) | Baseline, halfway and at the end of the intervention 18 weeks after the intervention, and at the 6 months follow up (42 weeks after baseline)
  The MHC-SF measures emotional, social and psychological wellbeing and is a self-report with 14 items
Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The PSQI is a self-report questionnaire that assesses sleep quality over a one-month interval and consists of 19 individual items.
Alcohol consumption and alcohol-related problems according to the Alcohol Use Disorders Identification test (AUDIT) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The AUDIT consists of 10 items scoring both consumption and alcohol-related problems. We will use the total scale on consumption and problem drinking
Treatment success according to the Outcome Questionnaire-45 | The questionnaire will be administered after every five modules of the intervention.
  a questionnaire to measure treatment success. It has three subscales: 1. Symptomatic distress (25 items, including symptoms of depression, anxiety and drug dependency, 2. Interpersonal relations (11 items) en 3. Social Role (9 items) .
Dietary intake of the participant according to a self devised questionnaire | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The questionnaire is a nutrition list with 25 items to measure the dietary intake of patients
Activity level defined as the daily number of steps | From baseline up to the 6 months follow up (42 weeks after baseline)
  The daily number of steps will be measured using the Fitbit Zip as described by Naslund et al., 2016
Body height of the participant as assessed by a stadiometer | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Body height in meters
Body weight of the participant as assessed by a medical weight scale | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Body weight in kilograms
Waist circumference of the participant as assessed using a tape meter line | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Waist circumference in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Cath, MD PhD, Principal Investigator — University Medical Center Groningen; Marjolein Berger, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - GGZ Drenthe, Assen, Drenthe
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ormel J, Von Korff M, Burger H, Scott K, Demyttenaere K, Huang YQ, Posada-Villa J, Pierre Lepine J, Angermeyer MC, Levinson D, de Girolamo G, Kawakami N, Karam E, Medina-Mora ME, Gureje O, Williams D, Haro JM, Bromet EJ, Alonso J, Kessler R. Mental disorders among persons with heart disease - results from World Mental Health surveys. Gen Hosp Psychiatry. 2007 Jul-Aug;29(4):325-34. doi: 10.1016/j.genhosppsych.2007.03.009. PMID 17591509
- [Background] Knol MJ, Heerdink ER, Egberts AC, Geerlings MI, Gorter KJ, Numans ME, Grobbee DE, Klungel OH, Burger H. Depressive symptoms in subjects with diagnosed and undiagnosed type 2 diabetes. Psychosom Med. 2007 May;69(4):300-5. doi: 10.1097/PSY.0b013e31805f48b9. Epub 2007 Apr 30. PMID 17470664